CLINICAL TRIAL: NCT00830089
Title: A Prospective Randomised Controlled Trial of the Efficacy of a Transversus Abdominis Plane Block in Laparoscopic Colorectal Surgery.
Brief Title: Trial of a Transversus Abdominis Plane (TAP) Block in Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09002
Record Dates: First submitted 2009-01-24; First posted 2009-01-27 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Post-operative Pain; Postoperative Nausea; Postoperative Complications
Keywords: Transversus abdominis plane block; Laparoscopic colorectal surgery; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications; Agnosia | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (Experimental): 40mls of 0.25% L-bupivicaine will be injected into the transversus abdominis plane (TAP) under ultrasound guidance - 20mls on either side of the abdomen.
  Interventions: Drug: Levobupivicaine 0.25%
- Standard care (No Intervention): No TAP block is given. Care is otherwise identical to arm 1

INTERVENTIONS:
Drug: Levobupivicaine 0.25% — 40mls of 0.25% L-bupivicaine will be injected into the transversus abdominis plane (TAP) under ultrasound guidance - 20mls on either side of the abdomen.
  Other Names: Chirocaine
  Arms: TAP block

SUMMARY:
Keyhole surgery for bowel disease has brought great benefits, enabling patients to recover quicker from surgery and so return to normal activities. Although keyhole surgery reduces pain following abdominal surgery, it still causes enough pain to require strong pain killing medications such as morphine-like drugs which, although good pain killers, can have a detrimental effect on the recovery of bowel function, leading to feelings of nausea and vomiting and ultimately delaying recovery. These side-effects can reduce the potential benefits from keyhole surgery and our "fast-track" recovery programmes.

The aim of this project is to assess the effectiveness of a new method of pain control after keyhole bowel surgery. The study involves the injection of local anaesthetic into the abdominal muscles once the patient is anaesthetised. Although use of local anaesthetic is common practice, we are looking at a new technique of injecting it called a transversus abdominis plane (or TAP) block. This technique will attempt to block the pain nerves to the abdomen prior to the operation beginning. We plan to investigate whether this new technique will reduce the amount of pain following keyhole bowel surgery. If successful, it might be used to further enhance people's recovery from bowel surgery.

DETAILED DESCRIPTION:
A considerable component of post-operative pain following abdominal surgery arises from the anterior abdominal wall. Although laparoscopic surgery has been shown to reduce post-operative pain scores compared to open surgery, there is still the problem of abdominal pain arising, in particular, from the specimen extraction site. Commonly used regimes to counter this pain include intravenous opiate-based patient-controlled analgesia (PCA) pumps, although such drugs can have a detrimental effect on the post-operative recovery of bowel function and leads to an increased risk of post-operative nausea and vomiting (PONV). The consequence of these gastrointestinal complications is that the benefits to patients of laparoscopic surgery with enhanced recovery programmes are not fully realised.

The benefits of adequate postoperative analgesia include a reduction in the postoperative stress response, reduction in postoperative morbidity, and in colorectal surgery, improved surgical outcome. Other benefits of effective regional analgesic techniques include reduced pain intensity, decrease incidence of side effects from analgesics (such as PONV), and improved patient comfort.

The innervation of the anterior abdominal wall comes from nerve afferents from T6-L1 running in the neurovascular plane which is found between internal oblique and transversus abdominis (TA). The transversus abdominis plane (TAP) block aims to block these nerves with local anaesthetic before they pierce the anterior abdominal wall. It has already shown to be effective in reducing pain in the first 24 hours after a laparotomy when compared to PCA with opiates and shown to have potential in a series of patients undergoing radical prostatectomy.

The potential improvement of this technique is weighed against the added risks of injecting into the neurovascular plane. There is a theoretical risk of a significant flank haematoma as a result of injury to the small vessels running with the nerves. In addition there is the small risk of inadvertent peritoneal puncture although the risk of any subsequent significant injury is very small and would likely be detected at the time of subsequent laparoscopy. Although there is one case report of a needle puncture to the liver due to previously unknown hepatomegaly, the injury was detected at laparotomy and the consequences were insignificant.

Experimental Methods and Design Patients would be randomised to receive either 20mls of local anaesthetic on each side of the abdomen in the TA plane or to receive no additional treatment. Both groups would receive local anaesthetic into the wounds at the end of the procedure. The TAP block would take place after induction of anaesthesia but before commencement of surgery. The TAP block would be carried out in a standardised manner using ultrasound guidance by two experienced anaesthetists with considerable experience in this technique. For blinding purposes, the site of entry on the skin for a TAP block will be covered with a plaster, irrespective of whether a block has been given.

A standardised anaesthetic and a standard post-operative analgesia regimen will be given to both groups.

Patients will be withdrawn from analysis if a colorectal resection does not take place or the surgery is converted to an open procedure, although data will continue to be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic colorectal resection at the Queen's Medical Centre, Nottingham

Exclusion Criteria:

* Known allergies to the local anaesthetic
* Any condition which may cause tolerance to opiates (eg chronic opioid use)
* Inability to use a PCA
* Patients less than 45kgs for whom local anaesthetic toxicity may become an issue
* Adults unable to consent for themselves

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Post-operative intravenous morphine use at 24 hours | 24 hours

SECONDARY OUTCOMES:
Pain score (visual analogue scale) | 24 hours
Nausea score | 24 hours
Length of stay | Days
Post-operative complications | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Austin Acheson, MD FRCS, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Walter CJ, Maxwell-Armstrong C, Pinkney TD, Conaghan PJ, Bedforth N, Gornall CB, Acheson AG. A randomised controlled trial of the efficacy of ultrasound-guided transversus abdominis plane (TAP) block in laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2366-72. doi: 10.1007/s00464-013-2791-0. Epub 2013 Feb 7. PMID 23389068